CLINICAL TRIAL: NCT02222272
Title: Effect of Prior Therapy With Nilotinib or Dasatinib on the Outcome After Allogeneic Stem Cell Transplantation for Patients With Chronic Myeloid Leukaemia
Brief Title: Effect of 2nd Gen TKI in CML
Status: Completed | Type: Observational
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: EBMT-42201038
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Myeloid Leukemia, Chronic
Keywords: cml; chronic myeloid leukemia; dasatinib; nilotinib; tki; second generation tki; 2nd generation tki
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Stem cell transplantation will continue to be a treatment option for patients with chronic myeloid leukaemia, despite the introduction of tyrosine kinase inhibitors. However, many patients will have received prior therapy with TKIs, including Nilotinib or Dasatinib at the time of allogeneic stem cell transplantation.

While the use of Imatinib prior to stem cell transplantation seems to have no adverse impact on the outcome of allogeneic stem cell transplantation little is known on the impact of prior use of second generation TK inhibitors.

Therefore this non interventional prospective study addresses this question and patients undergoing allogeneic stem cell transplantation after prior use of 2nd generation TKIs will be followed by the data office office on engraftment, treatment related mortality, relapse rate and survival, prospectively. Details on TKI therapy will be collected by the participating centers, retrospectively.

This is a non interventional prospective study. There is no upper limit to the number of patients entered, but it is estimated that up to 450 patients will be included in 150 centres for this non interventional prospective study. The registry will include patients for three years plus one more year for follow up and data analysis which should then be followed-up until the projected end of the non interventional prospective study.

DETAILED DESCRIPTION:
Chronic myeloid leukemia (CML) is a clonal disorder characterized by the chromosomal translocation t(9;22) which produces a fusion gene encoding the chimeric oncoprotein, BCR- ABL. This protein harbors a deregulated constitutive activated tyrosine kinase (TK) leading to leukemogenesis [1].

Imatinib mesylate, the first potent selective inhibitor of BCR-ABL TK [2] has become the frontline therapy for newly diagnosed CML patients [3]. It can induce haematologic and cytogenetic remission in all stages of CML, as well as in Ph positive acute lymphoblastic leukaemia (Ph+ ALL) with minimal toxicity [4, 5]. However, resistance and relapse during imatinib treatment are increasingly reported [6] and complete molecular remissions, as measured by polymerase chain reaction (PCR) are rare [7-9]. Loss of response to imatinib is frequently associated with mutations in the kinase domain of BCR-ABL which lead to impaired imatinib binding [10-12].

Nilotinib and Dasatinib are orally available kinase inhibitors that can overcome resistance to Imatinib [13 - 15]. Recent studies have demonstrated the efficacy and safety of both Nilotinib and Dasatinib in all stages of imatinib resistant CML. However, the long-term durability of these responses is uncertain yet, and substantial toxicity has been encountered [16]. Major adverse events observed during Nilotinib therapy were cytopenias, bone marrow suppression, gastrointestinal haemorrhage, diarrhea, cardiac dysfunction, liver toxicities and dermatitis [17-19] and during Dasatinib therapy grade 3/4 thrombocytopenia and neutropenia were reported in nearly half of the patients and non-hematologic toxicity consisted primarily of diarrhea, headache, fatigue, dyspnea and pleural effusion [20, 21].

Allogeneic stem cell transplantation (SCT) is now used mainly as salvage or curative therapy in patients with advanced CML who were previously treated with imatinib. While one study showed higher incidence of graft versus host disease (GVHD), venoocclusive disease (VOD) and transplant related mortality (TRM) [22], most studies have demonstrated that imatinib therapy prior to allogeneic SCT doesn't adversely affect transplantation outcome [23,24] . By contrast, previously used therapies for CML including busulfan and interferon alpha (if administrated less than 3 months before allogeneic SCT) have been reported to increase transplant related toxicities and mortality in CML patients undergoing allogeneic SCT [25, 26].

The impact of pre-transplant nilotinib or dasatinib therapy on transplant related complications, morbidity and outcome is mostly unknown and only two small case series have as yet been reported on this topic [27, 28]. However, allogeneic SCT will continue to be used as a salvage or curative therapy for CML especially in cases with resistance to kinase inhibitors or in patients at high risk of relapse, such as those in second chronic phase after blast crisis [29]. In the future 2nd generation TKIs may replace at least in part imatinib as frontline therapy for CML or will continue to be used in imatinib resistant patients. Nevertheless, in high risk patients allogeneic transplantation appears to remain the only curative treatment option.

For this reason, it is important to determine whether these novel treatments will not compromise transplantation outcome and increase transplant related complications.

Research design:

This is a non interventional prospective study with regard to SCT and follow-up. Patients agreeing to SCT will be identified from the EBMT database and from the transplant physicians. Transplant centres for the non interventional prospective study will be chosen from the EBMT centers that have transplanted patients with CML over the past 5 years. Transplant centers willing to participate will be registered with the EBMT Leiden Office. A prospective registry will keep record of all patients undergoing allogeneic SCT who had received prior treatment with 2nd generation TKIs and a specific data collection form (MED-B / MED-C) will be sent to the transplant centre to capture the relevant information at the appropriate intervals (day +100; 1 year; 2 years). Data will be collected regarding the safety and feasibility of stem cell transplant after Nilotinib or Dasatinib therapy (see endpoints).

The data on the treatment of patients with Nilotinib or Dasatinib before SCT will be collected retrospectively as part of the medical history (retrospective data collection). Participating centers planning an allogeneic SCT in a patient with CML previously treated with Nilotinib or Dasatinib will register the patient with the EBMT Leiden Office prior to transplant (day 0). A specific MED-C form will be sent to the centers immediately after registration.

All patients transplanted in an EBMT centre give specific consent for the collection and release of clinical data to the EBMT registry. Therefore, all patients registered in this non interventional prospective study would have signed an informed consent to authorise the release of medical information to the EBMT for the non interventional prospective study. Each centre will use their own standard consent form and information sheet. No specific consent form is envisaged for this non interventional prospective study.

Study Population:

This is an observational non interventional prospective study using the existing framework of the EBMT to identify and include patients. In 2006 560 patients with CML received an allotransplant, coming down from 800 in 2003. The percentage of patients transplanted not in first chronic phase is constantly increasing. Currently no data are available how many of those had previously been treated with 2nd generation TKI: it is however assumed, that also the number of patients transplanted after therapy with second generation TKI is increasing.

An estimate number is that for the next three years approximately 1500 allotransplants for CML will be done. 60% of these pts (n=900) would have received 2nd generation TKI. Assuming that at least 50% of them will be registered in the non interventional prospective study, it is expected that up to 450 patients will be identified over the next three years.

Patients response status to treatment with second line TKI (e.g. in stable CCyR, MCyR, or resistant to or progressing under 2nd line TKI) will be recorded to allow for identification of subgroups.

Research variables:

* Patients' features
* Centres' features
* Initial diagnosis
* Subclassification and status of disease at start 2nd generation TKI
* Response status to treatment with 2nd generation TKI prior to SCT
* TKI treatment (dose; duration; response)
* Subclassification and status of disease at HSCT
* Complications
* Additional therapies
* Relapse or progression
* Last disease and patient status
* Donor
* Transplantation
* Graft manipulation
* Engraftment
* Comorbid conditions
* Preparative treatment
* Graft versus Host disease
* Follow up

Data collection:

All correspondence will go through the data centre in Leiden. The data manager from the selected centre will complete the study forms. The data manager from the selected centre, national registry or the Paris office will collect the data forms and will enter the MED-B specific items. The MED-C items will be collected and entered by the data centre in Leiden. Data analysis will be done centrally at the CLWP office.

In case of inconsistencies a second check will be performed by a research assistant/data manager of the CLWP.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with chronic myeloid leukaemia in any phase (chronic, accelerated or blastic) who undergo allogeneic stem cell transplantation between 01/01/2010 and 30/09/2013 and have been previously treated with Nilotinib or Dasatinib, regardless of their response to these drugs.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: eligible patients from EBMT centres
Sampling Method: Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2014-03-19 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
non-relapse mortality (NRM) (treatment related mortality) | 1 year after HSCT

SECONDARY OUTCOMES:
treatment related toxic effects | 2 year after HSCT
overall survival | 2 years after HSCT
Event Free Survival | 2 years after HSCT
Relapse Rate | 2 years after HSCT

OTHER OUTCOMES:
outcome analyzed by response status to 2nd gen TKI prior to SCT | 2 year after HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schleuning, MD, Principal Investigator — Zentrum für Knochenmark und Blutstammzelltransplantation; Eduardo Olavarria, MD, Study Chair — Hospital de Navarra, Servicio de Hematologia, Pamplona, Spain; Nicolaus kroeger, MD, Study Chair — BMT Centre, University Hospital Eppendorf, Hamburg, Germany
Locations (10):
- Rigshospitalet, Copenhagen, Denmark
- Helsinki University Central Hospital, Helsinki, Finland
- Germany (2):
  - University of Freiburg, Freiburg im Breisgau
  - University of Muenster, Münster
- St Ivan & St Laszlo Hospital, Budapest, Hungary
- Chaim Sheba Medical Centre, Tel Litwinsky, Israel
- Medical University of Silesia, Katowice, Poland
- St Petersburg State Medical Pavlov University, Saint Petersburg, Russia
- King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia
- Hammersmith, London, United Kingdom